CLINICAL TRIAL: NCT00257101
Title: Stepped Intervention for Meds Adherence and Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 343; R01HL067439 (NIH)
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

INTERVENTIONS:
Behavioral: self-medication monitoring

SUMMARY:
To test the effectiveness of a stepped-care intervention involving 2 stages: (1) Self-Telemonitoring (STM) of blood pressure (BP) which uses a telephone transmission system (2) Telephone-Based Nurse Case Management (NCM), provided by a commercially available service.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The Medication Adherence and Blood Pressure Control Trial (ABC Trial) is a randomized controlled trial in a multicultural population of uncontrolled, hypertensive patients to test the effectiveness of a stepped-care intervention involving 2 stages: (1) Self-Telemonitoring (STM) of blood pressure (BP) which uses a telephone transmission system by which an easy-to-use modem, contained in the BP monitor, sends the BP measurements to a commercial service (Lifelink Monitoring) who then sends the measurements to the patient's health care provider; and (2) Telephone-Based Nurse Case Management (NCM), provided by a commercially available service (U-Med). The nurse case managers will call patients once/month, and provide counseling regarding BP control, and adherence to medication regimens. All patients in the intervention condition will begin with STM; after 3 months, patients whose BP has come under control remain in the STM condition; patients whose BP remain uncontrolled are then randomized, half to NCM + Self-Telemonitoring; the other half to continue in STM only (the design allows us to evaluate the effects of each arm of the intervention separately, and the combination; in addition, there will be a Usual Care condition). The focus is on an intervention strategy which readily transfers to a variety of usual health care situations. Both interventions are commercially available, and therefore are accessible to a wide range of health care providers, including smaller community-based clinics. An innovative aspect of the intervention is that the 2 commercial services will work together; the nurse case managers will receive BP reports from Lifelink, which the nurse will then use as a basis for counseling. The effectiveness of the interventions will be tested in 12 community-based clinics, which serve an economically disadvantaged, largely African American and Hispanic population, in New York City. The main outcome measures are medication adherence, determined by electronic drug event monitoring (MEMS), and pharmacy refill records, as well as BP control. Study duration is 1 year. The multilevel focus of the interventions is on provider as well as patient behavior. Reviews will be conducted for each patient at study discharge, recording data on clinic BP measurements during the previous 12 months, if any, doctor appointments, ER visits, medication changes, and evidence that the physician has responded to the interventions. The long-term goals of the research are to assess the medical and cost effectiveness of the interventions separately, and combined.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as hypertensive; chart data indicating poor BP control on two successive visits; pharmacy records indicate poorly adherence in previous 6 months
* Patients may have other co-morbid conditions
* On at least one antihypertensive medication
* Fluent in English or Spanish

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Gerin — Columbia University Health Sciences